CLINICAL TRIAL: NCT03733444
Title: A Phase 3, Randomized, Double-blind, Parallel-group, Placebo-controlled, Multi-center Study to Evaluate the Efficacy and Safety of Two Doses of GLPG1690 in Addition to Local Standard of Care for Minimum 52 Weeks in Subjects With Idiopathic Pulmonary Fibrosis
Brief Title: A Clinical Study to Test How Effective and Safe GLPG1690 is for Participants With Idiopathic Pulmonary Fibrosis (IPF) When Used Together With Standard of Care
Acronym: ISABELA2
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The benefit-risk profile no longer supports continuing the study
Sponsor: Galapagos NV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GLPG1690-CL-304; 2018-001406-29 (EudraCT Number)
Record Dates: First submitted 2018-11-05; First posted 2018-11-07 (Actual); Results first posted 2022-07-29 (Actual); Last update posted 2022-07-29 (Actual); Status verified 2022-07

CONDITIONS: Idiopathic Pulmonary Fibrosis
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis | interventions — GLPG1690

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- GLPG1690, 600 milligrams (mg) (Experimental): Participants received GLPG1690 (ziritaxestat) 600 mg as film-coated tablet orally, once daily (mean treatment duration was 332.9 days). Standard of care included either pirfenidone or nintedanib at a stable dose for at least 2 months before screening, and during screening; or neither pirfenidone or nintedanib (for any reason).
  Interventions: Drug: GLPG1690
- GLPG1690, 200 mg (Experimental): Participants received GLPG1690 (ziritaxestat) 200 mg as film-coated tablet orally, once daily (mean treatment duration was 336.9 days). Standard of care included either pirfenidone or nintedanib at a stable dose for at least 2 months before screening, and during screening; or neither pirfenidone or nintedanib (for any reason).
  Interventions: Drug: GLPG1690
- Placebo (Experimental): Participants received GLPG1690 (ziritaxestat) matching placebo tablets orally, once daily (mean treatment duration was 346.2 days). Standard of care included either pirfenidone or nintedanib at a stable dose for at least 2 months before screening, and during screening; or neither pirfenidone or nintedanib (for any reason).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GLPG1690 — GLPG1690, film-coated tablets for oral use.
  Other Names: ziritaxestat
  Arms: GLPG1690, 200 mg; GLPG1690, 600 milligrams (mg)
Drug: Placebo — Matching placebo, film-coated tablets for oral use.
  Arms: Placebo

SUMMARY:
The main purpose of this study was to see how GLPG1690 works together with the current standard treatment on your lung function and IPF disease in general. The study also investigated how well GLPG1690 is tolerated (for example if you get any side effects while on study drug).

ELIGIBILITY:
Inclusion Criteria:

* Male or female subject aged ≥40 years on the day of signing the Informed Consent Form (ICF).
* A diagnosis of IPF within 5 years prior to the screening visit, as per applicable American Thoracic Society (ATS)/European Respiratory Society (ERS)/Japanese Respiratory Society (JRS)/Latin American Thoracic Association (ALAT) guidelines at the time of diagnosis.
* Chest high-resolution computed tomography (HRCT) historically performed within 12 months prior to the screening visit and according to the minimum requirements for IPF diagnosis by central review based on subject's HRCT only (if no lung biopsy (LB) available), or based on both HRCT and LB (with application of the different criteria in either situation). If an evaluable HRCT <12 months prior to screening is not available, an HRCT can be performed at screening to determine eligibility, according to the same requirements as the historical HRCT.
* Subjects receiving local standard of care for the treatment of IPF, defined as either pirfenidone or nintedanib, at a stable dose for at least two months before screening, and during screening; or neither pirfenidone or nintedanib (for any reason). A stable dose is defined as the highest dose tolerated by the subject during those two months.
* The extent of fibrotic changes is greater than the extent of emphysema on the most recent HRCT scan (investigator-determined).
* Meeting all of the following criteria during the screening period: FVC ≥45% predicted of normal, Forced expiratory volume in 1 second (FEV1)/FVC ≥0.7, diffusing capacity of the lung for carbon monoxide (DLCO) corrected for Hb ≥30% predicted of normal.
* Estimated minimum life expectancy of at least 30 months for non IPF related disease in the opinion of the investigator.
* Male subjects and female subjects of childbearing potential agree to use highly effective contraception/preventive exposure measures from the time of first dose of investigational medicinal product (IMP) (for the male subject) or the signing of the ICF (for the female subject), during the study, and until 90 days (male) or 30 days (female) after the last dose of IMP.
* Able to walk at least 150 meters during the 6-Minute Walk Test (6MWT) at screening Visit 1; without having a contraindication to perform the 6MWT or without a condition putting the subject at risk of falling during the test (investigator's discretion). The use of a cane is allowed, the use of a stroller is not allowed at all for any condition. At Visit 2, for the oxygen titration test, resting oxygen saturation (SpO2) should be ≥88% with maximum 6 L O2/minute; during the walk, SpO2 should be ≥83% with 6 L O2/minute or ≥88% with 0, 2 or 4 L O2/minute.

Exclusion Criteria:

* History of malignancy within the past 5 years (except for carcinoma in situ of the uterine cervix, basal cell carcinoma of the skin that has been treated with no evidence of recurrence, prostate cancer that has been medically managed through active surveillance or watchful waiting, squamous cell carcinoma of the skin if fully resected, and Ductal Carcinoma In Situ).
* Clinically significant abnormalities detected on ECG of either rhythm or conduction, a QT interval corrected for heart rate using Fridericia's formula (QTcF) >450 ms, or a known long QT syndrome. Patients with implantable cardiovascular devices (e.g. pacemaker) affecting the QT interval time may be enrolled in the study based upon investigator judgment following cardiologist consultation if deemed necessary, and only after discussion with the medical monitor.
* Acute IPF exacerbation within 6 months prior to screening and/or during the screening period. The definition of an acute IPF exacerbation is as follows: Previous or concurrent diagnosis of IPF; Acute worsening or development of dyspnea typically < 1 month duration; Computed tomography with new bilateral ground-glass opacity and/or consolidation superimposed on a background pattern consistent with usual interstitial pneumonia pattern and deterioration not fully explained by cardiac failure or fluid overload.
* Lower respiratory tract infection requiring treatment within 4 weeks prior to screening and/or during the screening period.
* Interstitial lung disease associated with known primary diseases (e.g. sarcoidosis and amyloidosis), exposures (e.g. radiation, silica, asbestos, and coal dust), or drugs (e.g. amiodarone).
* Diagnosis of severe pulmonary hypertension (investigator determined).
* Unstable cardiovascular, pulmonary (other than IPF), or other disease within 6 months prior to screening or during the screening period (e.g. acute coronary disease, heart failure, and stroke).
* Had gastric perforation within 3 months prior to screening or during screening, and/or underwent major surgery within 3 months prior to screening, during screening or have major surgery planned during the study period.
* History of nintedanib-related increase in ALT and/or AST of >5 x upper limit of the normal range (ULN) and increased susceptibility to elevated LFT; moderate to severe hepatic impairment (Child-Pugh B or C) and/or abnormal liver function test (LFT) at screening, defined as aspartate aminotransferase (AST), and/or alanine aminotransferase (ALT), and/or total bilirubin ≥1.5 x upper limit of the normal range (ULN), and/or gamma glutamyl transferase (GGT) ≥3 x ULN. Retesting is allowed once for abnormal LFT.
* Abnormal renal function defined as estimated creatinine clearance, calculated according to Cockcroft-Gault calculation (CCr) <30 mL/min. Retesting is allowed once.
* Use of any of the following therapies within 4 weeks prior to screening and during the screening period, or planned during the study: warfarin, imatinib, ambrisentan, azathioprine, cyclophosphamide, cyclosporine A, bosentan, methotrexate, sildenafil (except for occasional use), prednisone at steady dose >10 mg/day or equivalent.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 781 (Actual)
Dates: Start 2018-11-05 (Actual); Primary Completion 2021-03-30 (Actual); Study Completion 2021-03-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Galapagos Study Director, Study Director — Galapagos NV
Locations (132):
- United States (36):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Arizona Pulmonary Specialists, Phoenix, Arizona
  - University of Arizona College of Medicine, Tucson, Arizona
  - Keck School of Medicine of USC, Los Angeles, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - UC Davis Medical Center, Sacramento, California
  - University of California, San Francisco Medical Center, San Francisco, California
  - St. Francis Medical Institute, Clearwater, Florida
  - University of Miami, Miami, Florida
  - Renstar Medical Research, Ocala, Florida
  - Central Florida Pulmonary Group PA, Orlando, Florida
  - Piedmont Healthcare, Atlanta, Georgia
  - Emory University, Atlanta, Georgia
  - University of Chicago Medical Center, Chicago, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - Brigham and Womens Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - University of Michigan Health System (UMHS), Ann Arbor, Michigan
  - Spectrum Health Medical Group, Grand Rapids, Michigan
  - University of Minnesota Medical Center, Minneapolis, Minnesota
  - Cardio Pulmonary Associates, Chesterfield, Missouri
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Atlantic Respiratory Institute, Summit, New Jersey
  - Lovelace Scientific Resources Inc, Albuquerque, New Mexico
  - Albany Medical Center, Albany, New York
  - Columbia University Medical Center, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Ohio State University, Columbus, Ohio
  - Mercy Health - St. Vincent Medical Center, Toledo, Ohio
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Temple Lung Center, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Medical University of South Carolina - PPDS, Charleston, South Carolina
  - University of Vermont, Burlington, Vermont
  - Inova Fairfax Hospital, Falls Church, Virginia
- Argentina (6):
  - Centro Médico Dra de Salvo, Buenos Aires
  - Hospital Privado Centro Médico de Córdoba, Córdoba
  - CEMER Centro Médico de Enfermedades Respiratorias, Florida
  - Hospital Zonal Especializado de Agudos y Crónicos Dr. Antonio A. Cetrangolo, Luján
  - Instituto de Investigaciones Clínicas Mar Del Plata, Mar del Plata
  - Fundacion Scherbovsky, Mendoza
- Canada (8):
  - South Health Campus, Calgary
  - Hôtel Dieu Du Centre Hospitalier de L'université de Montréal, Montreal
  - McGill University Health Centre Research Institute, Montreal
  - Institut Universitaire de Cardiologie et de Pneumologie, Québec
  - Toronto General Hospital, Toronto
  - Vancouver General Hospital, Vancouver
  - Pacific Lung Research Center, Vancouver
  - Dr Anil Dhar Professional Medicine Corporation, Windsor
- France (4):
  - Hôpital Nord AP-HM, Marseille
  - Centre Hospitalier Regional Universitaire Montpellier, Montpellier
  - Groupe Hospitalier Bichat Claude Bernard, Paris
  - CHU de Reims, Reims
- Germany (7):
  - Kliniken der Stadt Koln GmbH, Cologne
  - Ruhrlandklinik, Essen
  - Praxis Dr. med. Claus Keller, Frankfurt
  - Universitätsmedizin Greifswald Klinik und Poliklinik für Innere Medizin B, Greifswald
  - Pneumologisches Forschungsinstitut, Großhansdorf
  - Lungenfachklinik Immenhausen, Immenhausen
  - Krankenhaus Bethanien - Klinik für Pneumologie und Allergologie, Solingen
- Hungary (4):
  - Semmelweis Egyetem, Budapest
  - Veszprem Megyei Tudogyogyintezet, Farkasgyepű
  - Borsod-Abaúj-Zemplén Megyei Központi Kórház és Egyetemi Oktató Kórház, Miskolc
  - Tüdőgyógyintézet Törökbálint, Törökbálint
- Israel (6):
  - Barzilai Medical Center, Ashkelon
  - Lady Davis Carmel Medical Center, Haifa
  - Hadassah University Hospital Ein Kerem, Jerusalem
  - Meir Medical Center, Kfar Saba
  - Rabin Medical Center - PPDS, Petah Tikva
  - Kaplan Medical Center, Rehovot
- Italy (6):
  - Azienda Ospedaliero Universitaria Policlinico Vittorio Emanuele, Catania, Sicily
  - Azienda Ospedaliero Universitaria Ospedali Riuniti di Ancona-Umberto I G.M. Lancisi G. Salesi, Ancona
  - Presidio Ospedaliero GB Morgagni L Pierantoni, Forlì
  - Ospedale S. Giuseppe Multimedica, Milan
  - Università Cattolica Del S Cuore, Roma
  - Azienda Ospedaliera Universitaria Senese, Siena
- Japan (21):
  - National Hospital Organization Ibarakihigashi National Hospital, Naka, Ibaraki
  - Tenryu Hospital, Hamamatsu, Shizuoka
  - Juntendo University Hospital, Bunkyō City
  - National Hospital Organization Kyushu Medical Center, Fukuoka
  - Fukuoka University Hospital, Fukuoka
  - NHO Okinawa Hospital, Ginowan
  - Hamamatsu University School of Medicine, Hamamatsu
  - National Hospital Organization Himeji Medical Center, Himeji
  - Hiroshima Prefectural Hospital, Hiroshima
  - Kobe City Medical Center General Hospital, Hyōgo
  - Saiseikai Kumamoto Hospital, Kumamoto
  - Nagasaki University Hospital, Nagasaki
  - Nagoya University Hospital, Nagoya
  - Japanese Red Cross Okayama Hospital, Okayama
  - National Hospital Organization Kinki-Chuo Chest Medical Center, Sakai
  - Tohoku Medical and Pharmaceutical Hospital, Sendai
  - Tosei General Hospital, Seto
  - Tokyo Medical University Hospital, Shinjuku-Ku
  - Tokushima University Hospital, Tokushima
  - Center Hospital of the National Center for Global Health and Medicine, Tokyo
  - Kanagawa Cardiovascular and Respiratory Center, Yokohama
- Mexico (4):
  - Centro de Investigación Medico Biologica y de Terapia Avanzada S.C., Guadalajara
  - Instituto Nacional De Enfermedades (INER), Mexico City
  - Hospital Universitatorio Dr. Jose Eleuterio González, Monterrey
  - Unidad de Investigación Clínica En Medicina SC, Monterrey
- Netherlands (6):
  - VU Medisch Centrum, Amsterdam
  - OLVG locatie Oost, Amsterdam
  - Martini Ziekenhuis, Groningen
  - Zuyderland Medisch Centrum, Heerlen
  - St. Antonius Ziekenhuis, Nieuwegein
  - Erasmus MC, Rotterdam
- New Zealand (4):
  - Greenlane Clinical Centre, Auckland
  - NZ Respiratory & Sleep Institute, Auckland
  - Christchurch Hospital, Christchurch
  - Waikato Hospital, Hamilton
- Poland (8):
  - Centrum Medycyny Oddechowej Mroz sp. j., Bialystok
  - Uniwersyteckie Centrum Kliniczne - PPDS, Gdansk
  - PULMAG Arkadiusz Brodowski, Grzegorz Gasior S. C., Katowice
  - SP ZOZ Szpital Uniwersytecki w Krakowie, Krakow
  - GRAŻYNA JASIENIAK-PINIS ATOPIA Niepubliczny Zakład Opieki Zdrowotnej Poradnie Specjalistyczne, Krakow
  - SPZOZ Uniwersytecki Szpital Kliniczny nr 1 im Norberta Barlickiego Uniwersytetu Medycznego w Lodzi, Lodz
  - ETG Lublin, Lublin
  - ETG Warszawa, Warsaw
- South Africa (6):
  - Tygerberg Hospital, Cape Town
  - University of Cape Town Lung Institute (UCTLI), Cape Town
  - Dr Ismail Abdullah Private Practice, Cape Town
  - Ethekwini Hospital, Durban
  - Gateway Private Hospital, Durban
  - Milpark Hospital, Johannesburg
- South Korea (6):
  - Soon Chun Hyang University Hospital Bucheon, Bucheon-si, Gyeonggi-do
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Gachon University Gil Medical Center, Incheon
  - Asan Medical Center - PPDS, Seoul
  - Samsung Medical Center, Seoul
  - Soon Chun Hyang University Hospital Seoul, Seoul

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ford P, Kreuter M, Brown KK, Wuyts WA, Wijsenbeek M, Israel-Biet D, Hubbard R, Nathan SD, Nunes H, Penninckx B, Prasad N, Seghers I, Spagnolo P, Verbruggen N, Hirani N, Behr J, Kaner RJ, Maher TM. An adjudication algorithm for respiratory-related hospitalisation in idiopathic pulmonary fibrosis. ERJ Open Res. 2024 Jan 29;10(1):00636-2023. doi: 10.1183/23120541.00636-2023. eCollection 2024 Jan. PMID 38288082
- [Derived] Maher TM, Ford P, Brown KK, Costabel U, Cottin V, Danoff SK, Groenveld I, Helmer E, Jenkins RG, Milner J, Molenberghs G, Penninckx B, Randall MJ, Van Den Blink B, Fieuw A, Vandenrijn C, Rocak S, Seghers I, Shao L, Taneja A, Jentsch G, Watkins TR, Wuyts WA, Kreuter M, Verbruggen N, Prasad N, Wijsenbeek MS; ISABELA 1 and 2 Investigators. Ziritaxestat, a Novel Autotaxin Inhibitor, and Lung Function in Idiopathic Pulmonary Fibrosis: The ISABELA 1 and 2 Randomized Clinical Trials. JAMA. 2023 May 9;329(18):1567-1578. doi: 10.1001/jama.2023.5355. PMID 37159034
- [Derived] Deng X, Salgado-Polo F, Shao T, Xiao Z, Van R, Chen J, Rong J, Haider A, Shao Y, Josephson L, Perrakis A, Liang SH. Imaging Autotaxin In Vivo with 18F-Labeled Positron Emission Tomography Ligands. J Med Chem. 2021 Oct 28;64(20):15053-15068. doi: 10.1021/acs.jmedchem.1c00913. Epub 2021 Oct 18. PMID 34662125
- [Derived] Maher TM, Kreuter M, Lederer DJ, Brown KK, Wuyts W, Verbruggen N, Stutvoet S, Fieuw A, Ford P, Abi-Saab W, Wijsenbeek M. Rationale, design and objectives of two phase III, randomised, placebo-controlled studies of GLPG1690, a novel autotaxin inhibitor, in idiopathic pulmonary fibrosis (ISABELA 1 and 2). BMJ Open Respir Res. 2019 May 21;6(1):e000422. doi: 10.1136/bmjresp-2019-000422. eCollection 2019. PMID 31179008

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with a centrally confirmed diagnosis of idiopathic pulmonary fibrosis (IPF) were enrolled at 121 sites.
Pre-assignment Details: A total of 1431 participants were screened for the study, and 781 were randomized and 777 were treated.
Groups:
- GLPG1690, 600 mg: Participants received GLPG1690 (ziritaxestat) 600 mg as film-coated tablet orally, once daily (mean treatment duration was 332.9 days). Standard of care included either pirfenidone or nintedanib at a stable dose for at least 2 months before screening, and during screening; or neither pirfenidone or nintedanib (for any reason).
Period: Overall Study
Arm/Group | GLPG1690, 600 mg | GLPG1690, 200 mg | Placebo
Started | 260 | 262 | 259
Treated | 259 | 260 | 258
Completed | 0 | 0 | 0
Not Completed | 260 | 262 | 259
Not completed — Adverse Event | 8 | 10 | 5
Not completed — Death | 20 | 19 | 11
Not completed — Lost to Follow-up | 3 | 0 | 1
Not completed — Lack of Efficacy | 0 | 1 | 1
Not completed — Physician Decision | 2 | 1 | 0
Not completed — Protocol Violation | 2 | 1 | 0
Not completed — Protocol Specified Withdrawal Criteria Met | 1 | 1 | 2
Not completed — Study Terminated by Sponsor | 203 | 209 | 221
Not completed — Withdrawal by Subject | 19 | 18 | 16
Not completed — Miscellaneous | 1 | 0 | 1
Not completed — Not Treated | 1 | 2 | 1

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) consisted of all randomized participants who received at least 1 dose of investigation product (IP).
Groups:
- Total: Total of all reporting groups
Arm/Group | GLPG1690, 600 mg | GLPG1690, 200 mg | Placebo | Total
Number analyzed (Participants) | 259 | 260 | 258 | 777
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.2 (7.2) | 69.7 (7.3) | 70.6 (6.6) | 69.8 (7.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50 | 47 | 49 | 146
  Male | 209 | 213 | 209 | 631
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 32 | 34 | 28 | 94
  Not Hispanic or Latino | 217 | 215 | 218 | 650
  Unknown or Not Reported | 10 | 11 | 12 | 33
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 1 | 2 | 5
  Asian | 72 | 72 | 68 | 212
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1 | 2
  Black or African American | 2 | 0 | 1 | 3
  White | 174 | 178 | 178 | 530
  More than one race | 0 | 1 | 2 | 3
  Unknown or Not Reported | 8 | 8 | 6 | 22
Forced Vital Capacity [Mean (Standard Deviation); unit: Milliliter (mL)] — Forced vital capacity (FVC) (in milliliter [mL]) is the maximum amount of air exhaled from lungs by a participant after taking their deepest possible breath, as measured by spirometry. Population: FAS population with available data.
  Milliliter (mL)
    number analyzed (Participants) | 259 | 260 | 256 | 775
    (all) | 2775.66 (823.17) | 2768.63 (701.90) | 2749.54 (785.10) | 2764.67 (770.66)

OUTCOME MEASURES:

1. Primary Outcome: Annual Rate of Decline in Forced Vital Capacity (FVC) up to Week 52
Description: FVC (in mL) is the maximum amount of air exhaled from lungs by a participant after taking their deepest possible breath, as measured by spirometry.
Time Frame: Baseline up to week 52
Population: Full Analysis Set
Measure: Least Squares Mean (Standard Error); unit: mL/year
Arm/Group | GLPG1690, 600 mg | GLPG1690, 200 mg | Placebo
Number analyzed (Participants) | 259 | 260 | 258
mL/year | -173.8 (18.04) | -174.9 (17.65) | -176.6 (17.74)
Statistical Analysis 1: Comparison: GLPG1690, 600 mg vs Placebo; Test type: Superiority; p = 0.9123, Coefficient Regression Model — P-value was based on random coefficient regression model (linear slope model) on FVC values; Treatment effect was determined by using estimated slopes for each treatment group on basis of time-by-treatment interaction term from mixed model; Least Squares (LS) Mean difference = 2.8, 95% CI 2-sided [-46.9 to 52.4], Standard Error of Mean 25.29
Statistical Analysis 2: Comparison: GLPG1690, 200 mg vs Placebo; Test type: Superiority; p = 0.9456, Coefficient Regression Model — P-value was based on random coefficient regression model (linear slope model) on FVC values; [statistical method as in outcome 1, analysis 1]; LS Mean difference = 1.7, 95% CI 2-sided [-47.4 to 50.8], Standard Error of Mean 25.01

2. Secondary Outcome: Percentage of Participants With Disease Progression Up to 52 Weeks
Description: Disease progression was defined as the composite occurrence of more than or equal to (>=)10 percent (%) absolute decline in percent predicted forced vital capacity (%FVC) or all-cause mortality. FVC (in mL) is the maximum amount of air exhaled from lungs by a participant after taking their deepest possible breath, as measured by spirometry.
Time Frame: Up to week 52
Population: Full Analysis Set
Measure: Number; unit: Percentage of participants
Arm/Group | GLPG1690, 600 mg | GLPG1690, 200 mg | Placebo
Number analyzed (Participants) | 259 | 260 | 258
Percentage of participants | 23.9 | 23.1 | 22.1
Statistical Analysis 1: Comparison: GLPG1690, 600 mg vs Placebo; Test type: Superiority; p = 0.5162, Regression, Logistic; Odds Ratio (OR) = 1.15, 95% CI 2-sided [0.76 to 1.74]
Statistical Analysis 2: Comparison: GLPG1690, 200 mg vs Placebo; Test type: Superiority; p = 0.7566, Regression, Logistic; Odds Ratio (OR) = 1.07, 95% CI 2-sided [0.71 to 1.62]

3. Secondary Outcome: Percentage of Participants With Respiratory-Related Hospitalization Until End of Study (EoS)
Description: Percentage of participants with respiratory related to hospitalization were reported in this measure.
Time Frame: Up to EoS (week 125)
Population: Full Analysis Set
Measure: Number; unit: Percentage of participants
Arm/Group | GLPG1690, 600 mg | GLPG1690, 200 mg | Placebo
Number analyzed (Participants) | 259 | 260 | 258
Percentage of participants | 13.5 | 10.8 | 6.6
Statistical Analysis 1: Comparison: GLPG1690, 600 mg vs Placebo; Test type: Superiority; Hazard Ratio (HR) = 2.15, 95% CI 2-sided [1.20 to 3.85] — Hazard ratio and 95% confidence interval originated from a Cox proportional hazards model for time to first respiratory-related hospitalization
Statistical Analysis 2: Comparison: GLPG1690, 200 mg vs Placebo; Test type: Superiority; Hazard Ratio (HR) = 1.69, 95% CI 2-sided [0.93 to 3.10] — [estimate comment as in outcome 3, analysis 1]

4. Secondary Outcome: Change From Baseline in St.George's Respiratory Questionnaire (SGRQ) Total Score at Week 52
Description: SGRQ is a 50-item paper questionnaire designed to measure and quantify the impact of chronic respiratory disease on health-related quality of life (QOL) and well-being, split into 3 domains: symptoms score assessing the frequency and severity of respiratory symptoms (Items 1-8), activity score assessing the effects of breathlessness on mobility and physical activity (Items 11-17 and 36 to 44), and impacts score assessing the psychosocial impact of the disease (Items 9-10, 18-35 and 45-50). Each item has a specific weight.
  Domain scores = 100 * summed weights from positive items in that component/sum of maximum weights for all non-missing items in that component
  Total score = 100 * summed weights from positive items in the questionnaire/sum of maximum weights for all non-missing items in the questionnaire
  Scores were weighted such that each domain score ranged from 0 to 100 and the total score ranged from 0 to 100, with higher scores indicating the poorer health-related QOL.
Time Frame: Baseline, week 52
Population: Full Analysis Set
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | GLPG1690, 600 mg | GLPG1690, 200 mg | Placebo
Number analyzed (Participants) | 259 | 260 | 258
Score on a scale | 4.6 (1.13) | 4.3 (1.08) | 4.7 (1.10)
Statistical Analysis 1: Comparison: GLPG1690, 600 mg vs Placebo; Test type: Superiority; p = 0.9370, Mixed Models Analysis — LS mean difference (95% CI) per treatment group with treatment, time (categorical), treatment-by-time interaction, stratum and baseline SGRQ total score as fixed effects and participant as random effect; LS Mean difference = -0.1, 95% CI 2-sided [-3.2 to 3.0]
Statistical Analysis 2: Comparison: GLPG1690, 200 mg vs Placebo; Test type: Superiority; p = 0.8064, Mixed Models Analysis — [p-value comment as in outcome 4, analysis 1]; LS Mean difference = -0.4, 95% CI 2-sided [-3.4 to 2.7]

5. Secondary Outcome: Annual Rate of Decline of FVC Until EoS
Description: as for outcome 1
Time Frame: Baseline up to EoS (week 125)
Population: Full Analysis Set
Measure: Least Squares Mean (Standard Error); unit: mL/year
Arm/Group | GLPG1690, 600 mg | GLPG1690, 200 mg | Placebo
Number analyzed (Participants) | 259 | 260 | 258
mL/year | -179.5 (15.96) | -174.4 (15.63) | -182.4 (15.72)
Statistical Analysis 1: Comparison: GLPG1690, 600 mg vs Placebo; Test type: Superiority; LS Mean difference = 2.9, 95% CI 2-sided [-41.1 to 46.8], Standard Error of Mean 23.39 — The treatment effect was determined by using estimated slopes for each study group on the basis of the time-by-treatment interaction term from the mixed model
Statistical Analysis 2: Comparison: GLPG1690, 200 mg vs Placebo; Test type: Superiority; LS Mean difference = 8.0, 95% CI 2-sided [-35.5 to 51.5], Standard Error of Mean 22.16 — [estimate comment as in outcome 5, analysis 1]

6. Secondary Outcome: Percentage of Participants With Disease Progression Until EoS
Description: Disease progression was defined as the composite occurrence of >=10% absolute decline in percent predicted %FVC or all-cause mortality. FVC (in mL]) is the maximum amount of air exhaled from lungs by a participant after taking their deepest possible breath, as measured by spirometry.
Time Frame: Up to EoS (week 125)
Population: Full Analysis Set
Measure: Number; unit: Percentage of participants
Arm/Group | GLPG1690, 600 mg | GLPG1690, 200 mg | Placebo
Number analyzed (Participants) | 259 | 260 | 258
Percentage of participants | 31.7 | 27.7 | 26.7
Statistical Analysis 1: Comparison: GLPG1690, 600 mg vs Placebo; Test type: Superiority; Odds Ratio (OR) = 1.32, 95% CI 2-sided [0.90 to 1.94] — Odds ratio and 95% confidence interval originated from a logistic regression
Statistical Analysis 2: Comparison: GLPG1690, 200 mg vs Placebo; Test type: Superiority; Odds Ratio (OR) = 1.06, 95% CI 2-sided [0.72 to 1.56] — Odds ratio and 95% confidence interval originated from a logistic regression

7. Secondary Outcome: Change From Baseline in St. George's Respiratory Questionnaire (SGRQ) Total Score at Week 100
Description: as for outcome 4
Time Frame: Baseline, week 100
Population: Full Analysis Set
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | GLPG1690, 600 mg | GLPG1690, 200 mg | Placebo
Number analyzed (Participants) | 259 | 260 | 258
Score on a scale | 12.1 [3.0 to 21.2] | 14.8 [4.6 to 25.1] | 11.2 [1.6 to 20.8]
Statistical Analysis 1: Comparison: GLPG1690, 600 mg vs Placebo; Test type: Superiority; LS Mean difference = 0.9, 95% CI 2-sided [-12.4 to 14.1] — The treatment effect was determined by using estimated least square mean difference between each active treatment group and placebo from the mixed model
Statistical Analysis 2: Comparison: GLPG1690, 200 mg vs Placebo; Test type: Superiority; LS Mean difference = 3.6, 95% CI 2-sided [-10.4 to 17.6] — [estimate comment as in outcome 7, analysis 1]

8. Secondary Outcome: Percentage of Participants With All Cause Hospitalization Until EoS
Description: Percentage of participants with all cause hospitalization was reported for this measure.
Time Frame: Up to EoS (week 125)
Population: Full Analysis Set
Measure: Number; unit: Percentage of participants
Arm/Group | GLPG1690, 600 mg | GLPG1690, 200 mg | Placebo
Number analyzed (Participants) | 259 | 260 | 258
Percentage of participants | 20.8 | 18.8 | 14.0
Statistical Analysis 1: Comparison: GLPG1690, 600 mg vs Placebo; Test type: Superiority; Hazard Ratio (HR) = 1.54, 95% CI 2-sided [1.01 to 2.35] — Hazard ratio and 95% confidence interval originated from a Cox proportional hazards model for time to first all cause hospitalization
Statistical Analysis 2: Comparison: GLPG1690, 200 mg vs Placebo; Test type: Superiority; Hazard Ratio (HR) = 1.40, 95% CI 2-sided [0.91 to 2.16] — Hazard ratio and 95% confidence interval originated from a Cox proportional hazards model for time to all cause hospitalization

9. Secondary Outcome: Percentage of Participants With Respiratory Related Mortality Until EoS
Description: Percentage of participants with respiratory related mortality until end of study were reported for this study.
Time Frame: Up to EoS (week 125)
Population: Full Analysis Set
Measure: Number; unit: Percentage of participants
Arm/Group | GLPG1690, 600 mg | GLPG1690, 200 mg | Placebo
Number analyzed (Participants) | 259 | 260 | 258
Percentage of participants | 5.8 | 4.2 | 1.6

10. Secondary Outcome: Percentage of Participants Hospitalized for Non-Elective Lung Transplant Until EoS
Description: Percentage of Participants who were hospitalized for lung transplant were reported for this measure.
Time Frame: Up to EoS (week 125)
Population: Full Analysis Set
Measure: Number; unit: Percentage of participants
Arm/Group | GLPG1690, 600 mg | GLPG1690, 200 mg | Placebo
Number analyzed (Participants) | 259 | 260 | 258
Percentage of participants | 0 | 0 | 0

11. Secondary Outcome: Percentage of Participants With Acute Idiopathic Pulmonary Fibrosis (IPF) Exacerbation Until EoS
Description: Percentage of participants with acute IPF exacerbation until end of study were reported for this measure.
Time Frame: Up to EoS (week 125)
Population: Full Analysis Set
Measure: Number; unit: Percentage of participants
Arm/Group | GLPG1690, 600 mg | GLPG1690, 200 mg | Placebo
Number analyzed (Participants) | 259 | 260 | 258
Percentage of participants | 5.4 | 3.1 | 1.9
Statistical Analysis 1: Comparison: GLPG1690, 600 mg vs Placebo; Test type: Superiority; Hazard Ratio (HR) = 2.92, 95% CI 2-sided [1.04 to 8.14] — Hazard ratio and 95% confidence interval originated from a Cox proportional hazards model for time to first acute IPF exacerbation
Statistical Analysis 2: Comparison: GLPG1690, 200 mg vs Placebo; Test type: Superiority; Hazard Ratio (HR) = 1.68, 95% CI 2-sided [0.55 to 5.13] — [estimate comment as in outcome 11, analysis 1]

12. Secondary Outcome: Percentage of Participants With All Cause Mortality or Hospitalization for Non-elective Lung Transplant Until EoS
Description: Percentage of participants with all-cause mortality or hospitalization for non-elective lung transplant were reported for this measure.
Time Frame: Up to EoS (week 125)
Population: Full Analysis Set
Measure: Number; unit: Percentage of participants
Arm/Group | GLPG1690, 600 mg | GLPG1690, 200 mg | Placebo
Number analyzed (Participants) | 259 | 260 | 258
Percentage of participants | 8.1 | 6.9 | 3.9
Statistical Analysis 1: Comparison: GLPG1690, 600 mg vs Placebo; Test type: Superiority; Hazard Ratio (HR) = 2.27, 95% CI 2-sided [1.06 to 4.82] — Hazard ratio and 95% confidence interval originated from a Cox proportional hazards model for time to first all cause mortality or hospitalization for non-elective lung transplant
Statistical Analysis 2: Comparison: GLPG1690, 200 mg vs Placebo; Test type: Superiority; Hazard Ratio (HR) = 1.87, 95% CI 2-sided [0.86 to 4.06] — [estimate comment as in outcome 12, analysis 1]

13. Secondary Outcome: Percentage of Participants With All Cause Mortality, Hospitalization for Non-elective Lung Transplant or Hospitalization for Qualifying for Lung Transplant Until EoS
Description: Percentage of participants with all-cause mortality or hospitalization for qualifying for lung transplant were reported for this measure.
Time Frame: Up to EoS (week 125)
Population: Full Analysis Set
Measure: Number; unit: Percentage of participants
Arm/Group | GLPG1690, 600 mg | GLPG1690, 200 mg | Placebo
Number analyzed (Participants) | 259 | 260 | 258
Percentage of participants | 8.1 | 6.9 | 3.9
Statistical Analysis 1: Comparison: GLPG1690, 600 mg vs Placebo; Test type: Superiority; Hazard Ratio (HR) = 2.27, 95% CI 2-sided [1.06 to 4.82] — Hazard ratio and 95% confidence interval originated from a Cox proportional hazards model for time to first all cause mortality, hospitalization for non-elective lung transplant or hospitalization for qualifying for lung transplant
Statistical Analysis 2: Comparison: GLPG1690, 200 mg vs Placebo; Test type: Superiority; Hazard Ratio (HR) = 1.87, 95% CI 2-sided [0.86 to 4.06] — [estimate comment as in outcome 13, analysis 1]

14. Secondary Outcome: Percentage of Participants With All-Cause Mortality or Hospitalization That Meets >=10% Absolute Decline in %FVC or Respiratory-Related Hospitalization Until EoS
Description: Percentage of participants with all-cause mortality or respiratory related hospitalization that meets >=10% absolute decline in %FVC or respiratory-related hospitalization were reported for this measure.
Time Frame: Up to EoS (week 125)
Population: Full Analysis Set
Measure: Number; unit: Percentage of participants
Arm/Group | GLPG1690, 600 mg | GLPG1690, 200 mg | Placebo
Number analyzed (Participants) | 259 | 260 | 258
Percentage of participants | 16.6 | 12.7 | 8.9
Statistical Analysis 1: Comparison: GLPG1690, 600 mg vs Placebo; Test type: Superiority; Hazard Ratio (HR) = 1.99, 95% CI 2-sided [1.20 to 3.31] — Hazard ratio and 95% confidence interval originated from a Cox proportional hazards model for time to first all-cause mortality or hospitalization that meets >=10% absolute decline in %FVC or respiratory-related hospitalization
Statistical Analysis 2: Comparison: GLPG1690, 200 mg vs Placebo; Test type: Superiority; Hazard Ratio (HR) = 1.49, 95% CI 2-sided [0.88 to 2.54] — [estimate comment as in outcome 14, analysis 1]

15. Secondary Outcome: Percentage of Participants With All-Cause Mortality or Respiratory-Related Hospitalizations Until EoS
Description: Percentage of participants with all-cause mortality or respiratory related hospitalization were reported for this measure.
Time Frame: Up to EoS (week 125)
Population: Full Analysis Set
Measure: Number; unit: Percentage of participants
Arm/Group | GLPG1690, 600 mg | GLPG1690, 200 mg | Placebo
Number analyzed (Participants) | 259 | 260 | 258
Percentage of participants | 16.6 | 12.7 | 8.9
Statistical Analysis 1: Comparison: GLPG1690, 600 mg vs Placebo; Test type: Superiority; Hazard Ratio (HR) = 1.99, 95% CI 2-sided [1.20 to 3.31] — Hazard ratio and 95% confidence interval originated from a Cox proportional hazards model for time to first all-cause mortality or respiratory-related hospitalizations
Statistical Analysis 2: Comparison: GLPG1690, 200 mg vs Placebo; Test type: Superiority; Hazard Ratio (HR) = 1.49, 95% CI 2-sided [0.88 to 2.54] — [estimate comment as in outcome 15, analysis 1]

16. Secondary Outcome: FVC at Week 52
Description: as for outcome 1
Time Frame: Week 52
Population: FAS with available data at specified time point.
Measure: Mean (Standard Error); unit: mL
Arm/Group | GLPG1690, 600 mg | GLPG1690, 200 mg | Placebo
Number analyzed (Participants) | 127 | 137 | 131
mL | 2707.73 (66.096) | 2652.20 (61.173) | 2654.66 (73.437)

17. Secondary Outcome: Change From Baseline in FVC at Week 52
Description: as for outcome 1
Time Frame: Baseline, week 52
Population: FAS with available data at specified time point.
Measure: Mean (Standard Error); unit: mL
Arm/Group | GLPG1690, 600 mg | GLPG1690, 200 mg | Placebo
Number analyzed (Participants) | 127 | 137 | 131
mL | -153.78 (21.291) | -156.34 (17.410) | -177.39 (21.349)

18. Secondary Outcome: Percent Change From Baseline in FVC at Week 52
Description: as for outcome 1
Time Frame: Baseline, week 52
Population: FAS with available data at specified time point.
Measure: Mean (Standard Error); unit: Percent change
Arm/Group | GLPG1690, 600 mg | GLPG1690, 200 mg | Placebo
Number analyzed (Participants) | 127 | 137 | 131
Percent change | -5.71 (0.770) | -5.85 (0.690) | -6.42 (0.807)

19. Secondary Outcome: FVC at Week 100
Description: as for outcome 1
Time Frame: Week 100
Population: FAS with available data at specified time point.
Measure: Mean (Standard Error); unit: mL
Arm/Group | GLPG1690, 600 mg | GLPG1690, 200 mg | Placebo
Number analyzed (Participants) | 4 | 2 | 3
mL | 2474.0 (210.660) | 2897.50 (613.500) | 2937.67 (349.968)

20. Secondary Outcome: Change From Baseline in FVC at Week 100
Description: as for outcome 1
Time Frame: Baseline, week 100
Population: FAS with available data at specified time point.
Measure: Mean (Standard Error); unit: mL
Arm/Group | GLPG1690, 600 mg | GLPG1690, 200 mg | Placebo
Number analyzed (Participants) | 4 | 2 | 3
mL | -328.58 (123.456) | 134.0 (3.000) | -93.64 (321.208)

21. Secondary Outcome: Percent Change From Baseline in FVC at Week 100
Description: as for outcome 1
Time Frame: Baseline, week 100
Population: FAS with available data at specified time point.
Measure: Mean (Standard Error); unit: Percent change
Arm/Group | GLPG1690, 600 mg | GLPG1690, 200 mg | Placebo
Number analyzed (Participants) | 4 | 2 | 3
Percent change | -11.75 (4.481) | 5.07 (1.012) | -1.46 (11.279)

22. Secondary Outcome: Percentage of Participants With Absolute Categorical Change From Baseline in Percent FVC at Week 52: FVC Change Within ≤5
Description: as for outcome 1
Time Frame: Baseline, week 52
Population: FAS with available data at specified time point.
Measure: Number; unit: Percentage of participants
Arm/Group | GLPG1690, 600 mg | GLPG1690, 200 mg | Placebo
Number analyzed (Participants) | 127 | 137 | 131
Percentage of participants | 94.5 | 94.2 | 96.2

23. Secondary Outcome: Percentage of Participants With Absolute Categorical Change From Baseline in Percent FVC at Week 100: FVC Change Within ≤5
Description: as for outcome 1
Time Frame: Baseline, week 100
Population: FAS with available data at specified time point
Measure: Number; unit: Percentage of participants
Arm/Group | GLPG1690, 600 mg | GLPG1690, 200 mg | Placebo
Number analyzed (Participants) | 4 | 2 | 3
Percentage of participants | 100 | 100 | 66.7

24. Secondary Outcome: Percentage of Participants With Absolute Categorical Change From Baseline in Percent FVC at Week 52: FVC Change Within ≤10
Description: as for outcome 1
Time Frame: Baseline, week 52
Population: FAS with available data at specified time point.
Measure: Number; unit: Percentage of participants
Arm/Group | GLPG1690, 600 mg | GLPG1690, 200 mg | Placebo
Number analyzed (Participants) | 127 | 137 | 131
Percentage of participants | 98.4 | 100 | 99.2

25. Secondary Outcome: Percentage of Participants With Absolute Categorical Change From Baseline in Percent FVC at Week 100: FVC Change Within ≤10
Description: as for outcome 1
Time Frame: Baseline, week 100
Population: FAS with available data at specified time point.
Measure: Number; unit: Percentage of participants
Arm/Group | GLPG1690, 600 mg | GLPG1690, 200 mg | Placebo
Number analyzed (Participants) | 4 | 2 | 3
Percentage of participants | 100 | 100 | 66.7

26. Secondary Outcome: Percentage of Participants With Treatment Emergent Adverse Events (TEAEs) and Serious TEAEs
Description: Safety was assessed by adverse events (AEs), which included abnormalities identified during a medical test (e.g. laboratory tests, vital signs, electrocardiogram, etc.) if the abnormality induced clinical signs or symptoms, needed active intervention, interruption or discontinuation of study drug or was clinically significant. A Treatment emergent AE (TEAE) was defined as any AE that started or worsened after the first dose of study drug up to 30 days after the last dose of study drug. AEs were considered serious (SAEs) if the AE resulted in death, was life-threatening, resulted in persistent or significant disability/incapacity or substantial disruption of the ability to conduct normal life functions, resulted in congenital anomaly, or birth defect or required inpatient hospitalization or led to prolongation of hospitalization.
Time Frame: Baseline up to EoS (up to Week 125)
Population: Full Analysis Set
Measure: Number; unit: Percentage of participants
Arm/Group | GLPG1690, 600 mg | GLPG1690, 200 mg | Placebo
Number analyzed (Participants) | 259 | 260 | 258
Percentage of participants
  TEAE | 81.1 | 85.8 | 75.6
  Serious TEAE | 24.7 | 24.2 | 16.3

27. Secondary Outcome: Changes From Baseline in Leicester Cough Questionnaire (LCQ) Total Score and Individual Domain Score at Week 52 and Week 100
Description: Cough was evaluated using the LCQ. The LCQ is a 19-item questionnaire split into three domains: physical, psychological, and social. Scores were calculated by domain (range from 1 to 7) and then the total score was calculated by adding the individual domain score. Total score ranged from 3 to 21, with higher scores indicated a better health status.
Time Frame: Baseline, week 52, week 100
Population: FAS with available data at specified time point,
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | GLPG1690, 600 mg | GLPG1690, 200 mg | Placebo
Number analyzed (Participants) | 132 | 145 | 138
Score on a scale
  Physical score: Change at Week 52 | -0.187 (0.857) | -0.103 (0.925) | -0.219 (1.087)
  Physical score: Change at Week 100: number analyzed (Participants) | 10 | 8 | 9
  Physical score: Change at Week 100 | -0.463 (0.825) | -0.734 (1.141) | 0.000 (1.427)
  Psychological score: Change at Week 52 | -0.205 (1.004) | -0.040 (1.146) | -0.260 (1.215)
  Psychological score: Change at Week 100: number analyzed (Participants) | 10 | 8 | 9
  Psychological score: Change at Week 100 | -0.857 (1.313) | -0.518 (1.426) | 0.206 (1.136)
  Social score: Change at Week 52 | -0.178 (0.979) | -0.028 (1.122) | -0.232 (1.252)
  Social score: Change at Week 100: number analyzed (Participants) | 10 | 8 | 9
  Social score: Change at Week 100 | -0.450 (1.039) | -0.563 (1.406) | -0.139 (1.888)
  Total score: Change at Week 52 | -0.569 (2.606) | -0.171 (2.884) | -0.711 (3.291)
  Total score: Change at Week 100: number analyzed (Participants) | 10 | 8 | 9
  Total score: Change at Week 100 | -1.770 (3.038) | -1.815 (3.755) | 0.067 (3.999)

28. Secondary Outcome: Changes From Baseline in Visual Analogue Score (VAS): Cough at Week 52 and Week 100
Description: Cough was assessed using VAS score, ranged from 0 (no cough) to 100 millimeter (mm) (worst possible cough).
Time Frame: Baseline, week 52, week 100
Population: FAS with available data at specified time point.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | GLPG1690, 600 mg | GLPG1690, 200 mg | Placebo
Number analyzed (Participants) | 131 | 144 | 138
mm
  Change at Week 52 | 2.8 (26.4) | 2.8 (23.5) | 6.7 (28.9)
  Change at Week 100: number analyzed (Participants) | 10 | 8 | 9
  Change at Week 100 | 11.0 (34.0) | 14.0 (16.3) | -9.7 (18.0)

29. Secondary Outcome: Change From Baseline in Visual Analogue Score (VAS): Urge to Cough at Week 52 and Week 100
Description: Urge to Cough was assessed using VAS score, ranged from 0 (no urge to cough) to 100 mm (highest urge to cough).
Time Frame: Baseline, week 52, week 100
Population: FAS with available data at specified time point.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | GLPG1690, 600 mg | GLPG1690, 200 mg | Placebo
Number analyzed (Participants) | 131 | 144 | 138
mm
  Change at Week 52 | 4.8 (26.3) | 1.9 (25.9) | 6.7 (28.2)
  Change at Week 100: number analyzed (Participants) | 10 | 8 | 9
  Change at Week 100 | 8.7 (27.4) | 5.0 (17.1) | -15.8 (19.3)

30. Secondary Outcome: Changes From Baseline in EuroQOL 5-Dimensions Questionnaire at Week 52 and Week 100
Description: EuroQol outcome measurements was a printed 20 centimeter (cm) EQ visual analogue scale (EQ VAS) that appears somewhat like a thermometer, on which a score from 0 (worst imaginable health state or death) to 100 (best imaginable health state) was marked by the participant (or, when necessary, their proxy) with the scale in view.
Time Frame: Baseline, week 52, week 100
Population: FAS with available data at specified time point.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | GLPG1690, 600 mg | GLPG1690, 200 mg | Placebo
Number analyzed (Participants) | 133 | 146 | 139
Score on a scale
  Change at Week 52 | -5.9 (13.5) | -6.1 (15.3) | -3.7 (16.8)
  Change at Week 100: number analyzed (Participants) | 10 | 8 | 9
  Change at Week 100 | -11.2 (19.4) | -11.6 (20.1) | -4.7 (17.7)

31. Secondary Outcome: Changes From Baseline in King's Brief Interstitial Lung Disease (K-BILD) at Week 52 and Week 100
Description: The King's Brief Interstitial Lung Disease questionnaire (K-BILD) was specifically developed to analyze the health status of participants with OLD, the questionnaire consists of of 15 items (assessed by participants on scale ranging from 1 to 7, where 1 and 7 represents worst and best health status). Items are compiled into 3 domains: breathlessness and activities (range: 0-21), psychological (range: 0-34), and chest symptoms (range: 0-8). To score the K-BILD, the Likert response scale weightings for individual items are combined and scores are transformed to a range of 0-100 by using logit values (higher scores indicate better health status).
Time Frame: Baseline, week 52, week 100
Population: FAS with available data at specified time point.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | GLPG1690, 600 mg | GLPG1690, 200 mg | Placebo
Number analyzed (Participants) | 132 | 144 | 138
Score on a scale
  Breathlessness and Activities Score: Change at Week 52 | -2.876 (14.375) | -3.897 (13.668) | -2.414 (15.146)
  Breathlessness and Activities Score: Change at Week 100: number analyzed (Participants) | 10 | 8 | 9
  Breathlessness and Activities Score: Change at Week 100 | -8.530 (10.854) | -14.425 (12.995) | -1.411 (19.779)
  Psychological Score: Change at Week 52 | -3.508 (14.858) | -0.334 (16.875) | -1.769 (15.757)
  Psychological Score: Change at Week 100: number analyzed (Participants) | 10 | 8 | 9
  Psychological Score: Change at Week 100 | -4.170 (14.095) | 1.337 (22.141) | 0.778 (17.225)
  Chest Symptoms Score: Change at Week 52 | -4.213 (17.865) | -2.980 (17.775) | -5.159 (18.986)
  Chest Symptoms Score: Change at Week 100: number analyzed (Participants) | 10 | 8 | 9
  Chest Symptoms Score: Change at Week 100 | -4.760 (16.485) | -17.275 (21.758) | 4.333 (13.605)
  Total Score: Change at Week 52 | -2.241 (9.816) | -1.397 (10.030) | -2.009 (9.876)
  Total Score: Change at Week 100: number analyzed (Participants) | 10 | 8 | 9
  Total Score: Change at Week 100 | -5.080 (8.977) | -6.125 (14.278) | -0.156 (11.250)

32. Secondary Outcome: Area Under The Concentration Time Curve of Ziritaxtestat
Description: Area under the concentration time curve of ziritaxtestat was reported
Time Frame: Sparse samples collected on day 1 pre-dose, day 85 post-dose, day 237 post-dose, day 183 pre-dose, day 365 pre-dose
Population: Pharmacokinetic Analysis Set: All randomized participants who received at least one dose of IP and for whom evaluable PK data were available.
Measure: Median (90% Confidence Interval); unit: Nanogram * milliliter per hour (ng*mL/h)
Groups:
- GLPG1690, 200 mg: Participants received GLPG1690 (ziritaxestat) 200 mg as film-coated tablet orally, once daily (mean treatment duration was 336.9 days).
- GLPG1690, 600 mg: Participants received GLPG1690 (ziritaxestat) 600 mg as film-coated tablet orally, once daily (mean treatment duration was 332.9 days).
- GLPG1690 200 mg/Nintedanib: Participants received GLPG1690 (ziritaxestat) 200 mg, film-coated tablets orally once daily (mean GLPG1690 exposure was up to 325.3 days) in addition to local standard of care. Standard of care included nintedanib at a stable dose for at least 2 months before screening, and during screening;
- GLPG1690 600 mg/Nintedanib: Participants received GLPG1690 (ziritaxestat) 600 mg, film-coated tablets orally once daily (mean GLPG1690 exposure was up to 325.3 days) in addition to local standard of care. Standard of care included nintedanib at a stable dose for at least 2 months before screening, and during screening;
- GLPG1690 200 mg/Pirfenidone: Participants received GLPG1690 (ziritaxestat) 200 mg, film-coated tablets orally once daily (mean GLPG1690 exposure was up to 325.3 days) in addition to local standard of care. Standard of care included pirfenidone at a stable dose for at least 2 months before screening, and during screening;
- GLPG1690 600 mg/Pirfenidone: Participants received GLPG1690 (ziritaxestat) 600 mg, film-coated tablets orally once daily (mean GLPG1690 exposure was up to 325.3 days) in addition to local standard of care. Standard of care included pirfenidone at a stable dose for at least 2 months before screening, and during screening;
Arm/Group | GLPG1690, 200 mg | GLPG1690, 600 mg | GLPG1690 200 mg/Nintedanib | GLPG1690 600 mg/Nintedanib | GLPG1690 200 mg/Pirfenidone | GLPG1690 600 mg/Pirfenidone
Number analyzed (Participants) | 31 | 29 | 45 | 47 | 51 | 49
Nanogram * milliliter per hour (ng*mL/h) | 12058 [10935.81 to 13180.19] | 43640 [40056.29 to 47223.71] | 8006 [7210.62 to 8801.38] | 36135 [33155.43 to 39114.57] | 6570 [6022.87 to 7117.13] | 24777 [22452.09 to 27101.91]

33. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of Ziritaxtestat
Description: Maximum Observed Plasma Concentration of Ziritaxtestat was reported.
Time Frame: Sparse samples collected on day 1 pre-dose, day 85 post-dose, day 237 post-dose, day 183 pre-dose, day 365 pre-dose
Population: Pharmacokinetic Analysis Set
Measure: Median (90% Confidence Interval); unit: Nanogram per milliliter (ng/mL)
Groups:
- GLPG1690 200 mg/Nintedanib: Participants received GLPG1690 (ziritaxestat) 200 mg, film-coated tablets orally once daily (mean GLPG1690 exposure was up to 325.3 days) in addition to local standard of care. Standard of care included nintedanib at a stable dose for at least 2 months before screening, and during screening.
- GLPG1690 600 mg/Nintedanib: Participants received GLPG1690 (ziritaxestat) 600 mg, film-coated tablets orally once daily (mean GLPG1690 exposure was up to 325.3 days) in addition to local standard of care. Standard of care included nintedanib at a stable dose for at least 2 months before screening, and during screening.
- GLPG1690 200 mg/Pirfenidone: Participants received GLPG1690 (ziritaxestat) 200 mg, film-coated tablets orally once daily (mean GLPG1690 exposure was up to 325.3 days) in addition to local standard of care. Standard of care included pirfenidone at a stable dose for at least 2 months before screening, and during screening.
- GLPG1690 600 mg/Pirfenidone: Participants received GLPG1690 (ziritaxestat) 600 mg, film-coated tablets orally once daily (mean GLPG1690 exposure was up to 325.3 days) in addition to local standard of care. Standard of care included pirfenidone at a stable dose for at least 2 months before screening, and during screening.
Arm/Group | GLPG1690, 200 mg | GLPG1690, 600 mg | GLPG1690 200 mg/Nintedanib | GLPG1690 600 mg/Nintedanib | GLPG1690 200 mg/Pirfenidone | GLPG1690 600 mg/Pirfenidone
Number analyzed (Participants) | 31 | 29 | 45 | 47 | 51 | 49
Nanogram per milliliter (ng/mL) | 968 [902.25 to 1033.75] | 3529 [3315.25 to 3742.75] | 638 [591.23 to 684.77] | 2822 [2648.77 to 2995.23] | 606 [566.13 to 645.87] | 2280 [2111.2 to 2448.8]

34. Secondary Outcome: Change From Baseline in Functional Exercise Capacity, Assessed by The 6-Minute Walk Test (6MWT) Distance, at Week 52 and Week 100
Description: The 6MWT depicts the total distance covered by a participant during 6 minutes walking.
Time Frame: Baseline, week 52, week 100
Population: FAS with available data at specified time point.
Measure: Mean (Standard Error); unit: Meter
Arm/Group | GLPG1690, 600 mg | GLPG1690, 200 mg | Placebo
Number analyzed (Participants) | 101 | 107 | 108
Meter
  Change at Week 52 | -14.47 (6.610) | -36.33 (15.383) | -22.58 (6.128)
  Change at Week 100: number analyzed (Participants) | 0 | 0 | 1
  Change at Week 100 |  |  | -3.00

35. Secondary Outcome: Change From Baseline in Diffusing Capacity of Lung for Carbon Monoxide (DLCO) (Corrected for Hemoglobin [Hb]) at Week 52 and Week 100
Description: Change from baseline in diffusing capacity of the lung for carbon monoxide (percent predicted hemoglobin level corrected) was reported for this measure.
  mmol/min/kPa: Millimole per minute per kilopascal
Time Frame: Baseline, week 52 and week 100
Population: FAS with available data at specified time point.
Measure: Mean (Standard Error); unit: mmol/min/kPa
Arm/Group | GLPG1690, 600 mg | GLPG1690, 200 mg | Placebo
Number analyzed (Participants) | 97 | 111 | 104
mmol/min/kPa
  Change at week 52 | -0.307 (0.1004) | -0.247 (0.1019) | -0.394 (0.1104)
  Change at week 100: number analyzed (Participants) | 0 | 0 | 1
  Change at week 100 |  |  | -1.323

ADVERSE EVENTS:
Time Frame: Baseline up to 30 days after the last dose (Up to week 125)
Description: Full Analysis Set
Groups:
- Placebo: Participants received GLPG1690 (ziritaxestat) 600 mg as film-coated tablet orally, once daily (mean treatment duration was 332.9 days). Standard of care included either pirfenidone or nintedanib at a stable dose for at least 2 months before screening, and during screening; or neither pirfenidone or nintedanib (for any reason).
- GLPG1690, 600 mg: Participants received GLPG1690 (ziritaxestat) 200 mg as film-coated tablet orally, once daily (mean treatment duration was 336.9 days). Standard of care included either pirfenidone or nintedanib at a stable dose for at least 2 months before screening, and during screening; or neither pirfenidone or nintedanib (for any reason).
- GLPG1690, 200 mg: Participants received GLPG1690 (ziritaxestat) matching placebo tablets orally, once daily (mean treatment duration was 346.2 days). Standard of care included either pirfenidone or nintedanib at a stable dose for at least 2 months before screening, and during screening; or neither pirfenidone or nintedanib (for any reason).
Arm/Group | Placebo | GLPG1690, 600 mg | GLPG1690, 200 mg
All-Cause Mortality (participants affected / at risk) | 12/258 | 23/259 | 21/260
Serious Adverse Events (participants affected / at risk) | 42/258 | 64/259 | 63/260
Other Adverse Events (participants affected / at risk) | 117/258 | 141/259 | 134/260
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=258) | GLPG1690, 600 mg (N=259) | GLPG1690, 200 mg (N=260)
Peripheral artery stenosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Hypertensive emergency (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Peripheral artery thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Varicose vein (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (2)
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 2 (2)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0) | 0 (0)
Lung adenocarcinoma stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (3) | 0 (0) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Neoplasm prostate (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2) | 0 (0)
Oropharyngeal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (2)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Death (General disorders) | 1 (1) | 1 (1) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1)
Cystitis radiation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Lung diffusion test abnormal (Investigations) | 0 (0) | 0 (0) | 1 (1)
Oxygen saturation decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
SARS-CoV-2 test positive (Investigations) | 0 (0) | 0 (0) | 1 (1)
Scan myocardial perfusion abnormal (Investigations) | 0 (0) | 1 (1) | 0 (0)
Acute cardiac event (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 2 (2) | 2 (2) | 2 (3)
Angina unstable (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (2) | 0 (0)
Aortic valve stenosis (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiogenic shock (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure acute (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cor pulmonale (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
Coronary artery disease (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2)
Myocardial infarction (Cardiac disorders) | 2 (5) | 0 (0) | 2 (3)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Right ventricular failure (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Haemolytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (2) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Polycythaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (4)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (3) | 0 (0) | 2 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (3)
Eosinophilic pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Hypersensitivity pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Idiopathic pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 11 (15) | 20 (32) | 17 (24)
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 1 (2) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 7 (12) | 2 (2)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Cerebral infarction (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 2 (3) | 1 (1)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Parkinsonism (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 2 (3)
Glaucoma (Eye disorders) | 0 (0) | 0 (0) | 1 (2)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Duodenal ulcer perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Intestinal ischaemia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 (4) | 0 (0) | 0 (0)
Intestinal perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Sigmoid mesocolon hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2)
Drug-induced liver injury (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperplastic cholecystopathy (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (2)
Gallbladder cholesterolosis (Hepatobiliary disorders) | 0 (0) | 1 (2) | 0 (0)
Autoimmune nephritis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Glomerulonephritis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Renal cyst (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Renal colic (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Ureterolithiasis (Renal and urinary disorders) | 0 (0) | 1 (2) | 0 (0)
Renal vasculitis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Device failure (Product Issues) | 1 (1) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 0 (0)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (3)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 0 (0)
Cachexia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 4 (7) | 4 (9)
Bronchopulmonary aspergillosis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
COVID-19 pneumonia (Infections and infestations) | 1 (1) | 1 (2) | 2 (4)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Erysipelas (Infections and infestations) | 0 (0) | 0 (0) | 1 (2)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Peritonitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Liver abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Pneumonia (Infections and infestations) | 2 (4) | 6 (11) | 5 (5)
Pneumonia influenzal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 1 (2) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (2)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 2 (2) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 2 (2) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=258) | GLPG1690, 600 mg (N=259) | GLPG1690, 200 mg (N=260)
Weight decreased (Investigations) | 8 (9) | 14 (16) | 9 (14)
Cough (Respiratory, thoracic and mediastinal disorders) | 22 (27) | 24 (32) | 20 (23)
Idiopathic pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 14 (17) | 24 (34) | 18 (21)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 22 (25) | 14 (14) | 12 (14)
Headache (Nervous system disorders) | 15 (16) | 16 (19) | 14 (17)
Diarrhoea (Gastrointestinal disorders) | 47 (89) | 74 (199) | 58 (104)
Nausea (Gastrointestinal disorders) | 13 (14) | 23 (36) | 16 (22)
Back pain (Musculoskeletal and connective tissue disorders) | 6 (6) | 13 (14) | 6 (7)
Decreased appetite (Metabolism and nutrition disorders) | 9 (11) | 20 (23) | 14 (19)
Bronchitis (Infections and infestations) | 4 (9) | 14 (18) | 11 (17)
Nasopharyngitis (Infections and infestations) | 13 (14) | 16 (19) | 16 (22)
Upper respiratory tract infection (Infections and infestations) | 17 (22) | 18 (24) | 21 (24)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor must review and approve any results of the study or abstracts for professional meetings prepared by the investigator(s). Published data must not compromise the objectives of the study. Data from individual study centers in multicenter studies must not be published separately.

DOCUMENTS (2):
  • Study Protocol (2020-06-08): https://cdn.clinicaltrials.gov/large-docs/44/NCT03733444/Prot_000.pdf
  • Statistical Analysis Plan (2021-03-25): https://cdn.clinicaltrials.gov/large-docs/44/NCT03733444/SAP_001.pdf